CLINICAL TRIAL: NCT00273546
Title: A Randomized Phase III Multicenter Trial of Neoadjuvant Docetaxel (Taxotere®) Plus Cisplatin and 5-Fluorouracil (TPF) Versus Neoadjuvant Cisplatin Plus 5-Fluorouracil Followed by Concomitant Chemoradiotherapy to Improve the Overall Survival and Progression Free Survival in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Induction Chemotherapy Comparing Taxotere® Cisplatin and 5-Fluorouracil (TPF) With Standard Cisplatin and 5-Fluorouracil (PF) Followed by Chemoradiation in Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6043; RP-56976-V-324; NCT00004214 (obsolete NCT alias)
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cancer
Keywords: Head and Neck Cancer; Induction; Chemotherapy; Chemoradiotherapy
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: XRP6976 (Docetaxel/Taxotere)

SUMMARY:
* 1.To compare overall survival after treatment with the test tri-therapy (TPF: docetaxel plus cisplatin and 5FU) or the control treatment (PF: cisplatin plus 5-FU) followed by chemoradiotherapy in patients with locally advanced SCCHN.
* 2.The main secondary endpoint is progression free survival (PFS). The other secondary endpoints are to evaluate and compare improvement of local symptoms; time-to-treatment failure; quality of life; clinical complete response rate (CR and CR/PR); toxicity and to evaluate the relationship of tumor markers and response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically or cytologically proven squamous cell carcinoma of the head/neck.
* 2.Primary tumor sites eligible: oral cavity, oropharynx, hypopharynx, larynx. Although they are admittedly of squamous cell types, the following tumors will be excluded because their responsiveness to chemotherapy may differ: nasal, paranasal cavities; nasopharynx.
* 3.Stage 3 or 4 disease without evidence of distant metastases verified with Chest X-Ray, abdominal ultrasound or CT (liver function test abnormalities); bone scan in case of local symptoms.
* 4.At least one uni or bidimensionally measurable lesion.
* 5.Tumor considered as inoperable after evaluation by a multidisciplinary team (surgeon, medical oncologist and radiation oncologist). Criteria include : Technical unresectablility-ie tumor fixation/invasion to base of the skull or cervical vertebrae involvement of the nasopharynx and fixed lymph nodes; Physician's decision based on low surgical curability which includes all T3-4 stages, all N2-3 stages excluding T1N2; organ preservation.
* 6.No previous chemotherapy or radiotherapy for any reason and no previous surgery for SCCHN (other than biopsy) are allowed at time of study entry.
* 7.Age ³ 18 years.
* 8.WHO performance status of 0-1
* 9.No active alcohol addiction
* 10.Life expectancy ³ 12 weeks
* 11.Signed informed consent prior to beginning protocol specific procedures
* 12.Adequate bone marrow, hepatic and renal functions as evidenced by the following: Hematology (Bone Marrow): Neutrophil count ³ 2.0 x 10 9/L; Platelet count ³ 100 X 10 9/L; Hemoglobin ³ 10g/dL; Hepatic function : Total bilirubin WNL; ASAT (SGOT) and ALAT (SGPT) £ 2.5 X ULN; Alkaline phosphatase £ 5 X ULN; patients with ASAT or ALAT > 1.5 x ULN associated with alkaline phosphatase > 2.5 x ULN are not eligible for the study; Renal function: the creatinine clearance ³ 60 ml/min (actual or calculated by the Cockcroft-Gault method as follows: Weight (kg) X (140-age)/K x serum creatinine.
* 13.Patients must be available for treatment and follow up. Patients registered on this trial must be treated and followed at the participating center.

Exclusion Criteria:

* 1.Pregnant or lactating women or women of childbearing potential not using adequate contraception.
* 2.Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years. Any prior treatment with radiotherapy or chemotherapy is an exclusion criterion.
* 3.Symptomatic peripheral neuropathy ³ grade 2 by NCIC-CTG criteria.
* 4.Symptomatic altered hearing > grade 2 by NCIC-CTG criteria.
* 5.Other serious illnesses or medical conditions including but no limited to: Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry; History of significant neurologic or psychiatric disorders including dementia or seizures; Active uncontrolled infection; Active peptic ulcer; Hypercalcemia; Chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry.
* 6.Patients requiring intravenous alimentation.
* 7.Patients who experienced a weight loss of more than 20% of their body weight in the 3 months preceding study entry.
* 8.Concurrent treatment with any other anticancer therapy
* 9.Participation in an investigational trial within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 1999-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Overall survival after treatment with the test tri-therapy (TPF: docetaxel plus cisplatin and 5-FU) or the control treatment (PF: Cisplatin plus 5-FU) followed by chemoradiotherapy.

SECONDARY OUTCOMES:
The main secondary outcome is progression free survival (PFS).
The other secondary endpoints are improvement of local symptoms;time-to-treatment failure;quality of life;
clinical complete response rate (CR) and overall response rate(PR+CR) after chemotherapy and after locoregional therapy(chemoradiotherapy);
duration of response(CR and CR+PR); toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Study Chair — Dana-Farber Cancer Institute
Locations (6):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia

REFERENCES:
- [Result] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Derived] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014